CLINICAL TRIAL: NCT07056062
Title: Effect of Oral Calcium Carbonate on Uterine Contractility and Labor Outcomes: A Randomized Controlled Trial
Brief Title: Oral Calcium Supplementation in Labor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Arrowhead Regional Medical Center (Other)
Responsible Party: Principal Investigator, Tina Bui, MFM Fellow, Arrowhead Regional Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-16
Record Dates: First submitted 2025-06-21; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Uterine Contraction; Labor Complication; Labor Active Dilated Cm; Labor Dystocia; Labor Duration; Labor; Labor Delivery
Keywords: calcium carbonate; labor; vaginal delivery; cesarean delivery
MeSH Terms: conditions — Obstetric Labor Complications; Dystocia | interventions — Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group received a single oral dose of 2,000 mg calcium carbonate, consisting of four over-the-counter antacid tablets. This dose is well below the recommended daily maximum of 8,000 mg. The control group received no medication. Common side effects of calcium carbonate include constipation, bloating, and abdominal discomfort, while serious side effects such as hypercalcemia are rare.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of care (No Intervention): Received no medications but monitored for the duration of the study
- Calcium carbonate (Experimental): 2,000 mg PO calcium carbonate as a single dose
  Interventions: Drug: Calcium carbonate

INTERVENTIONS:
Drug: Calcium carbonate — 2,000 mg PO calcium carbonate as a single dose
  Other Names: TUMS
  Arms: Calcium carbonate

SUMMARY:
The goal of this clinical trial is to learn if oral calcium carbonate can improve uterine contractions and labor outcomes in term pregnancies. It will also evaluate the safety of calcium carbonate when used during labor. The main questions it aims to answer are:

Does oral calcium carbonate increase uterine contraction strength? Does it lead to shorter labor duration or higher vaginal delivery rates? What side effects or complications, if any, occur with calcium carbonate use during labor?

Researchers will compare oral calcium carbonate to no treatment to see if it helps improve labor efficiency and reduce cesarean delivery rates.

Participants will:

Be randomly assigned to receive either 2,000 mg of oral calcium carbonate or no intervention Undergo monitoring with an intrauterine pressure catheter to measure contraction strength Be observed for two hours without oxytocin to assess calcium's direct effect on contractions Have data collected on labor progression, delivery outcomes, and neonatal health

DETAILED DESCRIPTION:
In the United States, nearly one-third of deliveries are performed via cesarean section, with labor dystocia remaining a leading indication. Labor dystocia may result from a variety of maternal and fetal factors, including malposition, cephalopelvic disproportion, or ineffective uterine contractions. When contractions are inadequate, the standard intervention is intravenous oxytocin. However, prolonged or high-dose oxytocin administration can lead to receptor desensitization, reducing its effectiveness and increasing the risk of postpartum hemorrhage.

Calcium plays a key role in myometrial contractility by facilitating calcium influx through L-type channels in myometrial cells, which triggers intracellular calcium release and action potentials. During labor, upregulation of calcium channels enhances the uterus's responsiveness to contractile stimuli. Elevated serum calcium levels have been associated with stronger and more effective contractions.

Adjunctive intravenous calcium administration with oxytocin has been shown to improve labor outcomes, including higher rates of vaginal delivery within 24 hours of induction and reduce blood loss in cesarean deliveries. However, the potential role of oral calcium supplementation in enhancing labor progression has not been evaluated in clinical trials. Given its physiological relevance, accessibility, and low-risk profile, oral calcium may represent a simple adjunct to improve labor efficiency and reduce cesarean rates.

This study aims to evaluate the impact of oral calcium carbonate supplementation during labor on uterine contractility and clinical outcomes. The investigators hypothesize that calcium carbonate administered intrapartum will enhance uterine contractions, resulting in higher vaginal delivery rates, shorter time to delivery, and reduced blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Had an intrauterine pressure catheter in place
* Term gestation, greater than or equal to 37 weeks of gestation
* Singleton pregnancy
* Cephalic presentation
* > 18 years of age

Exclusion Criteria:

* incarceration
* multiple gestation
* active illicit drug use
* abnormal clinical pelvimetry
* Suspected fetal macrosomia defined as estimated fetal weight ≥4250 grams
* intrauterine growth restriction
* abnormal placentation
* prior cesarean delivery
* maternal history of arrhythmia
* hyperparathyroidism
* heart failure
* renal or hepatic failure
* nephrolithiasis
* receipt of medications known to affect uterine contractility-such as magnesium sulfate, terbutaline, or recent misoprostol in the last four hours

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Contraction Frequency | Two hours after receiving the study medication or, for control participants, two hours after enrollment.
  Recording the number of contractions in a ten-minute period for 2 hours
Uterine contraction strength | Two hours after receiving the study medication or, for control participants, two hours after enrollment.
  Recording Montevideo units every 30 minutes for 2 hours
Peak strength | Two hours after receiving the study medication or, for control participants, two hours after enrollment.
  Recording the max pressure generated during a contraction using an intrauterine pressure catheter during the 2-hour study period

SECONDARY OUTCOMES:
Duration of the first stage of labor | Calculated at the time of delivery
  Record the length of the first stage of labor from 6 cm to 10 cm dilation
Duration of the second stage of labor | Calculated at the time of delivery
  Record the time from 10 cm to delivery of the baby
Mode of delivery | Calculated at the time of delivery
  Determine whether or not patient had a spontaneous vaginal bleeding, operative vaginal delivery, or cesarean delivery
Pitocin dose | Calculated at the time of delivery
  Record the maximum dose of Pitocin used during labor
Postpartum hemorrhage | at the time of discharge (assessed up to 5 days)
  Determine which patients had a blood loss of greater than or equal to 1000 mL
Neonatal outcomes | at the time of discharge (assessed up to 5 days)
  Determine which babies were admitted to neonatal intensive care unit (NICU) and had a low 5- minute APGAR score

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Valenzuela, MD, Principal Investigator — Arrowhead Regional Medical Center
Locations (1):
- Arrowhead Regional Medical Center, Colton, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study has already been completed, will analyze data first and then decide

REFERENCES:
- [Background] Cai R, Chen L, Xing Y, Deng Y, Li J, Guo F, Liu L, Xie C, Yang J. RETRACTED: Oxytocin with calcium vs oxytocin for induction of labor in women with term premature rupture of membranes: a randomized controlled trial. Am J Obstet Gynecol MFM. 2024 Nov;6(11):101502. doi: 10.1016/j.ajogmf.2024.101502. Epub 2024 Sep 20. PMID 39307241
- [Background] Ansari JR, Yarmosh A, Michel G, Lyell D, Hedlin H, Cornfield DN, Carvalho B, Bateman BT. Intravenous Calcium to Decrease Blood Loss During Intrapartum Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2024 Jan 1;143(1):104-112. doi: 10.1097/AOG.0000000000005441. Epub 2023 Nov 3. PMID 37917943
- [Background] Papandreou L, Chasiotis G, Seferiadis K, Thanasoulias NC, Dousias V, Tsanadis G, Stefos T. Calcium levels during the initiation of labor. Eur J Obstet Gynecol Reprod Biol. 2004 Jul 15;115(1):17-22. doi: 10.1016/j.ejogrb.2003.11.032. PMID 15223159
- [Background] Pehlivanoglu B, Bayrak S, Dogan M. A close look at the contraction and relaxation of the myometrium; the role of calcium. J Turk Ger Gynecol Assoc. 2013 Dec 1;14(4):230-4. doi: 10.5152/jtgga.2013.67763. eCollection 2013. PMID 24592112
- [Background] Wray S, Jones K, Kupittayanant S, Li Y, Matthew A, Monir-Bishty E, Noble K, Pierce SJ, Quenby S, Shmygol AV. Calcium signaling and uterine contractility. J Soc Gynecol Investig. 2003 Jul;10(5):252-64. doi: 10.1016/s1071-5576(03)00089-3. PMID 12853086
- [Background] Obstetric care consensus no. 1: safe prevention of the primary cesarean delivery. Obstet Gynecol. 2014 Mar;123(3):693-711. doi: 10.1097/01.AOG.0000444441.04111.1d. PMID 24553167
- See also: Related Info — https://institutionalrepository.aah.org/cgi/viewcontent.cgi?article=2010&context=jpcrr
- See also: Related Info — https://www.researchgate.net/publication/331250259_Correlation_of_Calcium_Levels_With_The_Strenght_of_Uterus_Contraction_on_The_Active_Phase_of_First_Stage_Labor

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT07056062/Prot_SAP_ICF_000.pdf